CLINICAL TRIAL: NCT01823107
Title: Meso BioMatrix Acellular Peritoneum Matrix Breast Reconstruction Feasibility Trial
Brief Title: Feasibility Study of Meso BioMatrix Device for Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kensey Nash Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MESO-001
Record Dates: First submitted 2013-03-26; First posted 2013-04-04 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Meso BioMatrix; Breast; Breast Cancer; Mastectomy; Biologic Mesh; Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Meso BioMatrix Device (Experimental): All subjects will have the Meso BioMatrix device implanted along with a tissue expander during the first stage of breast reconstruction. During the second stage of breast reconstruction, the tissue expander is replaced with a breast implant.
  Interventions: Device: Meso BioMatrix Device

INTERVENTIONS:
Device: Meso BioMatrix Device

SUMMARY:
The purpose of the study is to evaluate the safety and feasibility of the use of Meso BioMatrix Acellular Peritoneum Matrix for the reinforcement of weakened soft tissue during 2-stage, tissue expander assisted breast reconstruction.

DETAILED DESCRIPTION:
Following mastectomy, women may elect to have breast reconstruction with autologous tissue or breast implants. Two-stage, tissue expander assisted breast reconstruction is one of the common surgical methods that could be selected to reconstruct the breast. This method either begins immediately after mastectomy (known as immediate breast reconstruction) or at some time afterward (known as delayed breast reconstruction). Historically, surgeons placed a tissue expander followed by the breast implant either completely or partially under the pectoralis muscle. However, this method of breast reconstruction has been associated with less favorable aesthetic outcomes.

Recently, surgeons started adding a surgical mesh derived from human cadaver skin during breast reconstruction procedures. In summary, during the first stage of the breast reconstruction, the plastic surgeon releases the pectoralis muscle from the chest wall. The surgeon then attaches the surgical mesh to the pectoralis muscle and to the chest wall just below the breast. This is done to create a pocket for the tissue expander. The tissue expander is implanted in the pocket and partially inflated. The tissue expander is gradually filled with saline over several weeks or months. Once the desired breast volume has been achieved, the second stage of the reconstruction takes place. In the second stage, the tissue expander is removed and replaced with a permanent saline or silicone gel breast implant.

Use of the human cadaver skin surgical mesh during breast reconstruction has been associated with less pain, fewer tissue expansion visits and improved aesthetic outcomes. However, the human cadaver skin surgical mesh adds significant cost to the procedure and some surgeons have reported an increased rate of post-operative complications.

Over the last 10 years, a number of surgical mesh devices have been cleared by the U.S. Food & Drug Administration (FDA) for the reinforcement and repair weak soft tissue or became available as tissue grafts from human donors. Some surgeons have published their experience with a number of these surgical mesh devices for breast reconstruction. However, at present, no surgical mesh device is approved or cleared by the FDA for use in breast reconstruction.

The Meso BioMatrix device was recently cleared by the FDA for reinforcement and repair of weak soft tissue. It is a surgical mesh device that is made from pig peritoneum, the tissue that lines the abdominal cavity. The tissue is thoroughly cleaned and sterilized before use. When implanted, the Meso BioMatrix device provides structural and mechanical support to weak soft tissue during the healing process.

This clinical trial is a feasibility trial. A feasibility trial is a clinical trial in which a device is being studied in a small group of people for a new use. Since the Meso BioMatrix device is not cleared specifically for use in breast reconstruction, it is considered investigational and must be studied in a controlled, step-wise series of clinical trials. Therefore, the results of this trial, if successful, may be used to design a larger clinical trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker
* Undergoing unilateral or bilateral, two-stage, tissue expander-assisted breast reconstruction
* Life expectancy greater than 18 months
* Agreement to return for the trial required follow-up visits

Exclusion Criteria:

* Body mass index ≥ 35
* Prior reconstructive breast surgery, breast augmentation, mastopexy or reduction mammoplasty
* History of chronic corticosteroid use
* Type I Diabetes
* History of radiation therapy to the chest
* Pre-operative treatment with induction chemotherapy for breast cancer
* Pregnancy
* Participating in another investigational drug or device trial that has not completed the follow-up period

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Forde Hansell, Study Director — DSM Biomedical
Locations (6):
- United States (6):
  - Henry Ford Health System, Detroit, Michigan
  - Long Island Plasic Surgical Group, PC, Garden City, New York
  - Long Island Plastic Surgical Group, PC, Garden City, New York
  - Cancer Center of America at Eastern Regional Medical Center / Dr. Glat Plastic & Reconstructive Surgery, Bala-Cynwyd, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah (Huntsman Cancer Hospital), Salt Lake City, Utah

REFERENCES:
- [Derived] Simpson AM, Higdon KK, Kilgo MS, Tepper DG, Alizadeh K, Glat PM, Agarwal JP. Porcine Acellular Peritoneal Matrix in Immediate Breast Reconstruction: A Multicenter, Prospective, Single-Arm Trial. Plast Reconstr Surg. 2019 Jan;143(1):10e-21e. doi: 10.1097/PRS.0000000000005095. PMID 30589773

RESULTS

PARTICIPANT FLOW:
Groups:
- Meso BioMatrix Acellular Peritoneum Matrix: All subjects had the Meso BioMatrix Acellular Peritoneum Matrix implanted along with a tissue expander during the first stage of breast reconstruction. After tissue expansion, the tissue expander was replaced with a breast implant during the second stage of reconstruction.
Period: Overall Study
Arm/Group | Meso BioMatrix Acellular Peritoneum Matrix
Started | 25
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Meso BioMatrix Acellular Peritoneum Matrix
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.0 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Breast Related Adverse Events
Description: Investigators evaluated each subject and each reconstructed breast for the occurrence of an adverse event from the first stage of reconstruction through the final follow-up visit. A breast related adverse event was defined as any untoward medical occurrence related to a reconstructed breast.
Time Frame: 18 months
Measure: Number; unit: Reconstructed breasts affected
Units Other Than Participants: Reconstructed breasts
Arm/Group | Meso BioMatrix Acellular Peritoneum Matrix
Number analyzed (Participants) | 25
Number analyzed (Reconstructed breasts) | 44
Reconstructed breasts affected | 12

2. Secondary Outcome: Measurement of Aesthetic Satisfaction With the Use of the Breast-Q Survey
Description: Subjects completed the reconstructive module of the BREAST-Q, a standardized instrument measuring patient satisfaction and health-related quality of life on a scale of 1 to 100, with higher scores indicating higher satisfaction. Completed Breast-Q questionnaires were scored according to the author's instructions. Aesthetic satisfaction was measured using the Breast-Q Satisfaction with Breasts subscale score.
Time Frame: 18 months (12 months after second stage reconstruction)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meso BioMatrix Acellular Peritoneum Matrix
Number analyzed (Participants) | 24
score on a scale | 71.2 (15.5)

3. Secondary Outcome: Rate of Reconstruction Failure
Description: Reconstruction failure was defined as a serious adverse event in a reconstructed breast resulting in unplanned removal of the prosthesis and/or Meso BioMatrix Acellular Peritoneum Matrix.
Time Frame: 18 months
Population: Forty-four (44) breasts were reconstructed among the 25 enrolled subjects. Reconstruction failure was evaluated on a per reconstructed breast basis.
Measure: Number; unit: Reconstructed breasts affected
Units Other Than Participants: Reconstructed breasts
Arm/Group | Meso BioMatrix Acellular Peritoneum Matrix
Number analyzed (Participants) | 25
Number analyzed (Reconstructed breasts) | 44
Reconstructed breasts affected | 3

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Meso BioMatrix Acellular Peritoneum Matrix
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 7/25
Other Adverse Events (participants affected / at risk) | 10/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Meso BioMatrix Acellular Peritoneum Matrix (N=25)
Seroma (Reproductive system and breast disorders) | 1
Fever (General disorders) | 1
Wound dehiscence (Reproductive system and breast disorders) | 4
Hematoma (Blood and lymphatic system disorders) | 1
Skin flap necrosis (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Meso BioMatrix Acellular Peritoneum Matrix (N=25)
Breast pain (Reproductive system and breast disorders) | 3
Skin rash (Skin and subcutaneous tissue disorders) | 3
Erythema (Respiratory, thoracic and mediastinal disorders) | 4

LIMITATIONS AND CAVEATS:
The trial allowed investigator discretion for perioperative medical management, including antibiotic administration, tissue expansion protocol, surgical drain placement, and drain duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT01823107/Prot_SAP_000.pdf